CLINICAL TRIAL: NCT01682590
Title: Impact on Mortality of the Timing of Renal Replacement Therapy in Patients With Severe Acute Kidney Injury in Septic Shock: the IDEAL-ICU Study (Initiation of Dialysis Early Versus Delayed in the Intensive Care Unit): Study Protocol for a Randomized Controlled Trial
Brief Title: I.D.E.A.L.-I.C.U. (Initiation of Dialysis EArly Versus deLayed in Intensive Care Unit)
Acronym: IDEAL-ICU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Quenot IDEAL-ICU
Record Dates: First submitted 2012-09-10; First posted 2012-09-11 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock; Acute Renal Failure (as Defined by the "Failure" Stage of the RIFLE Classification)
Keywords: septic shock; acute renal failure; renal remplacement therapy; mortality; intensive care; critical care; acute kidney injury
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: To investigate whether early initiation of RRT (within 12 hours after a diagnosis of acute renal insufficiency at the"failure" stage according to the RIFLE Criteria), will reduce 90-day mortality as compared to deferred initiation of RRT(48 to 60 hours after diagnosis), in intensive care unit (ICU) patients with septic shock who develop acute renal failure
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early initiation of RRT (Experimental): Start of RRT within a maximum of 12 hours after randomisation.
  Interventions: Procedure: Renal Remplacement Therapy
- Deferred RRT (Active Comparator): Start of RRT between 48 and 60 hours after randomisation.
  Interventions: Procedure: Renal Remplacement Therapy

INTERVENTIONS:
Procedure: Renal Remplacement Therapy — Investigators of each center will have the choice of the RRT technique based on their usual practice: intermittent hemodialysis, intermittent hemodiafiltration, continuous hemodialysis, continuous hemofiltration, continuous hemodiafiltration (typically the continuous techniques in the acute phase, followed by intermittent techniques after stabilization).
  In case of life threatening conditions within the 48 hours after randomisation (hyperkalemia, metabolic acidosis or pulmonary edema) the RRT will be initiated as soon as possible.
  In case of improvement of renal function within the 48 hours after randomisation (defined as the return of spontaneous urine output > 1000ml/24 hr or >2000ml/24hr with diuretics), RRT is not mandatory.

SUMMARY:
The purpose of this multicentric, randomized controlled trial is to assess whether the timing of renal replacement therapy initiation (early vs delayed) has an impact on mortality at 90 days in patients with severe acute kidney injury at the failure stage (according to RIFLE criteria) during the initial phase of septic shock.

DETAILED DESCRIPTION:
Acute renal failure is one of the most feared complications of septic shock and occurs in 51% of patients with these conditions. Mortality at 3 months ranges from 36% to 60%. To date, these exists no consensus regarding the optimal time to initiate renal remplacement therapy (RRT). Retrospective and observational studies have suggested that early initiation of RRT could help to improve prognosis in these patients. Therefore, we aim to investigate wether early initiation of RRT (within 12 hours after a diagnosis of acute renal insufficiency at the "failure" stage according to the RIFLE Criteria), will reduce 90-day mortality as compared to deferred initiation of RRT (48 to 60 hours after diagnosis), in intensive care unit (ICU) patients with septic shock who develop acute renal failure.

Secondary objectives include: to compare the impact of the two RRT strategies on 28, 180 et 360 day mortality, duration of mechanical ventilation, duration of RRT, duration of ICU stay and duration of overall hospital stay. In addition, quality of life at 90 and 360 days will be evaluated using the EQ5D questionnaire. Tolerance of both strategies will be compared in terms of metabolic disorders, arrhythmias, pulmonary oedema by overload, hypotension, hemorrhagic complications, and dependence on RRT at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

Adults (males or females, age >18 years) with septic shock who develop acute renal failure (as defined by the "Failure" stage of the RIFLE classification) will be eligible for inclusion.

Septic shock is defined as severe sepsis with at least 2 to 4 "SIRS" criteria and persistent hypotension despite adequate vascular filling and need vaso-active drugs.

SIRS is defined as the simultaneous presence of at least 2 of the following criteria :

* Body temperature ≥ 38°C ou ≤ 36°C
* Heart rate ≥ 90 bpm
* Respiratory rate ≥ 20/mn or PaCO2 ≤ 32 mmHg
* Leucocytes ≥ 12,000/mm3 or ≤ 4,000/mm3 or >10% immature forms.

Acute renal insufficiency is defined as the "failure" stage of the RIFLE classification, i.e. the presence of at least one of the following criteria:

* Increased creatinine x 3 times the baseline value
* Oliguria < 0.3 ml/kg/h for 12 hours
* Anuria (diuresis < 100ml) for at least 12 hours

All patients are required to provide informed consent after having been appropriately informed about the study. In case of temporary incapacity of the patient to sign, the consent form can be signed by a surrogate.

Exclusion Criteria:

Patients presenting any of the following criteria will not be eligible for inclusion in the study:

1. Patients with chronic renal at dialysis.
2. Patients presenting acute renal failure of type obstructive and patients already presenting emergency criteria for immediate hemodialysis at the time of randomization (i.e. hyperkalemia >6.5 mmol/L or pH<7.15 or pulmonary oedema by fluid overload)
3. Patients already had hemodialysis before their arrival in the intensive care unit
4. Pregnant women.
5. Moribund patients whose life expectancy is less than 24 hours
6. Patients unlikely to survive to 28 days because of uncontrollable comorbidities (e.g. cardiac, pulmonary or hepatic disease at the terminal stage, hepatorenal syndrome, uncontrolled cancer, severe post-anorexic encephalopathy…)
7. Patients with advance directives indicating their wish not to be resuscitated.
8. Patients under legal guardianship.
9. Patients participing in another interventional study that may influence the prognosis of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-07; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 90 days
  To investigate whether early initiation of RRT (within 12 hours after a diagnosis of acute renal insufficiency at the "failure" stage according to the RIFLE Criteria), will reduce 90-day mortality as compared to deferred initiation of RRT (48 to 60 hours after diagnosis), in intensive care unit (ICU) patients with septic shock who develop acute renal failure.

SECONDARY OUTCOMES:
Comparison of the tolerance and evaluation quality of life | 90 days
  Secondary objectives include: to compare the impact of the two RRT strategies on 28, 180 and 360 day mortality, duration of mechanical ventilation, duration of RRT, duration of ICU stay and duration of overall hospital stay. In addition, quality of life at 90 and 360 days will be evaluated using the EQ5D questionnaire. Tolerance of both strategies will be compared in terms of metabolic disorders, arrhythmias, pulmonary oedema by overload, hypotension, hemorrhagic complications, and dependence on RRT at hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre QUENOT, Study Director — Centre Hospitalier Universitaire Dijon; Saber Davide BARBAR, Principal Investigator — CHU de Nimes
Locations (27):
- France (27):
  - CH Avignon, Avignon
  - CH Belfort, Belfort
  - CHU Besançon, Besançon
  - CH de BOURG-EN-BRESSE, Bourg-en-Bresse
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Dieppe, Dieppe
  - CHU Dijon, Dijon
  - CH Sud Essonne - Site Etampes, Étampes
  - Hôpital Raymond-Poincaré GARCHES (AP-HP), Garches
  - CHU Grenoble, Grenoble
  - CH de LA ROCHE sur YON, La Roche-sur-Yon
  - Groupe Hospitalier de l'institut Catholique de LILLE, Lille
  - CHU de Lyon, Lyon
  - CHU Montpellier, Montpellier
  - CHU Lapeyronie, Montpellier
  - CHG Mulhouse, Mulhouse
  - CHU Nancy Brabois, Nancy
  - CHU Nîmes, Nîmes
  - CHR d'Orléans, Orléans
  - Hôpital Cochin, Paris
  - HOPITAL BICHAT Claude-Bernard, Paris
  - CH Périgueux, Périgueux
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Strasbourg - Nouvel hôpital civil, Strasbourg
  - CHR Metz, Thionville
  - CHRU Tours, Tours

REFERENCES:
- [Background] Barbar SD, Binquet C, Monchi M, Bruyere R, Quenot JP. Impact on mortality of the timing of renal replacement therapy in patients with severe acute kidney injury in septic shock: the IDEAL-ICU study (initiation of dialysis early versus delayed in the intensive care unit): study protocol for a randomized controlled trial. Trials. 2014 Jul 7;15:270. doi: 10.1186/1745-6215-15-270. PMID 24998258
- [Result] Barbar SD, Clere-Jehl R, Bourredjem A, Hernu R, Montini F, Bruyere R, Lebert C, Bohe J, Badie J, Eraldi JP, Rigaud JP, Levy B, Siami S, Louis G, Bouadma L, Constantin JM, Mercier E, Klouche K, du Cheyron D, Piton G, Annane D, Jaber S, van der Linden T, Blasco G, Mira JP, Schwebel C, Chimot L, Guiot P, Nay MA, Meziani F, Helms J, Roger C, Louart B, Trusson R, Dargent A, Binquet C, Quenot JP; IDEAL-ICU Trial Investigators and the CRICS TRIGGERSEP Network. Timing of Renal-Replacement Therapy in Patients with Acute Kidney Injury and Sepsis. N Engl J Med. 2018 Oct 11;379(15):1431-1442. doi: 10.1056/NEJMoa1803213. PMID 30304656
- [Result] Barbar SD, Dargent A, Quenot JP. Timing of Renal-Replacement Therapy in Acute Kidney Injury and Sepsis. N Engl J Med. 2019 Jan 24;380(4):399. doi: 10.1056/NEJMc1815142. No abstract available. PMID 30673539
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787